CLINICAL TRIAL: NCT04657913
Title: The Effect of Spray Use on Mouth Dryness and Thirst of Patients Undergone Major Abdominal Surgery: A Randomized Controlled Study
Brief Title: Mouth Dryness and Thirst of Patients Undergone Major Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Bediye Oztas, Principal investigator, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ankara Medipol University
Record Dates: First submitted 2020-09-28; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-09

CONDITIONS: Xerostomia; Thirst
Keywords: mouth dryness; thirst; saliva; oral health; major abdominal surgery; randomized controlled health
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cold water spray group (Experimental): application of cold water in the form of a spray to mouth of patients will be applied 2 times per hour, starting 2 hours after the end of the operation.
  Interventions: Other: cold water spray application
- cold saline spray group (Experimental): application of cold 0.9% SF (saline) in the form of a spray to mouth of patients will be applied 2 times per hour, starting 2 hours after the end of the operation.
  Interventions: Other: cold saline spray application
- control group (No Intervention): no intervention

INTERVENTIONS:
Other: cold water spray application — It will be sprayed into the mouth of patients every hour.
  Other Names: cold water spray
  Arms: cold water spray group
Other: cold saline spray application — It will be sprayed into the mouth of patients every hour.
  Other Names: cold saline spray
  Arms: cold saline spray group

SUMMARY:
The purpose of this study is to determine the effects of spray use on dry mouth and thirst of patients who had undergone major abdominal surgery. The methods used to alleviate the thirst and dry mouth experienced by patients undergoing major abdominal surgery are limited. This research was conducted as a randomized controlled trial.

DETAILED DESCRIPTION:
The study sample includes patients who had undergone major abdominal surgery induced by upper or lower gastrointestinal system malignancies. The patients who met the inclusion criteria were informed about the purpose of the study and were invited to the study. Those who accepted to participate in the study were included in the study.

Patients who had undergone major abdominal surgery with general anesthesia (induced by upper or lower gastrointestinal system malignancies), who do not have any oral and nasal diseases, who do not have visual, hearing, speech and understanding problems, who were in the American Society of Anesthesiologists (ASA) I and II grades, who were aged 18 or over and agreed to participate in the study were included.

Patients whose mouth and tongue mucosa integrity was degraded, who had a cognitive disorder, or were suffering from neurological, renal, cardiac or pulmonary disorders that could affect the test results, or who use psychoactive drugs were excluded.

The standard anesthesia protocol was implemented to all patients suitable for the study. In the postoperative period, the standard rational dose antibiotic therapy (1st generation cephalosporin + metronidazole), metoclopramide HCL, NSAIDs, LMWH, N-acetylcysteine (NAC), H2-receptor blockers (ranitidine HCL), pethidine HCL 50 mg/ml, when required, and maintenance fluid therapy (Combination of normal saline, lactated Ringer's and Dextrose) by their weight were administered to the patients.

First Control Group: No intervention was performed on the patients in the control group. To prevent ethical violations, patients received routine clinical practice (a small amount of water was administered orally, using a syringe).

Second Intervention Group: Cold water kept at +40 C in the refrigerator was added into 50cc spray-head bottles and administered to patients orally in the postoperative phase, by spraying twice hourly.

Third intervention Group: Cold normal saline (0.9% NaCl) kept at +40 C in the refrigerator was added into 50cc spray-head bottles and administered to patients orally in the postoperative phase, by spraying twice hourly.

No intervention was performed on patients from midnight thru 06:00 AM, in order not to disturb the circadian rhythms of all patients.

Considering surgery end time and circadian rhythms of patients, the data of the patients were recorded at the post-operative 4, 8, 20, 24, 36, 40th hours. The flow chart of the study is shown in Figure 1. In the cold water and cold normal saline applications, 50cc glass bottles, plastic spray head, and cover were used. New material was used for each patient.

Preoperative measurements: Patients' data such as age, gender, comorbid diseases, ASA (American Society of Anesthesiologists) grade, diagnosis, preoperative thirst intensity, preoperative mouth dryness intensity, preoperative oral health condition were recorded.

Outcome measurements Postoperative evaluations were made after the interventions. Intensity of Thirst: VAS with a range of 0-10 points (0: mild, 10 very severe) was used while the thirsty severity of all patients were evaluated.

Intensity of Mouth Dryness: VAS with a range of 0-10 points (0: never experiencing mouth dryness, 10: experiencing very intense mouth dryness) was used while the mouth dryness severity of all patients were evaluated.

Oral Health Condition: To assess patients' oral health condition, the Oral Health Assessment Tool (OHAT) was used. The first four items of the scale that assess lips, tongue, gums and tissue, and saliva were used. The lowest score to be obtained from the scale is 0, while the highest score is 8 (0=healthy; 1=changes; 2=unhealthy). A higher OHAT score indicates a poor oral condition.

Saliva PH: To measure the PH of saliva, the patient's saliva sample in a sterile container was assessed using PH test strips.

Patient Satisfaction: To evaluate patient satisfaction, overall satisfaction was scored using a 10-point numerical rating scale (NRS) from 0 (complete dissatisfaction) to 10 (complete satisfaction).

At the postoperative 4th hour, the severity of thirst and dry mouth, oral health status and saliva PH values were evaluated in terms of differences between the groups.

At the postoperative 8th hour, the severity of thirst and dry mouth, oral health status and saliva PH values were evaluated in terms of differences between the groups.

At the postoperative 20,24,36 and 40th hour, the severity of thirst and dry mouth, oral health status and saliva PH values were evaluated in terms of differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent major abdominal surgery under general anesthesia (due to lower and upper gastrointestinal tract malignancy)
* patients without oral and nasal disease
* patients who do not have vision, hearing, speech and understanding problems
* patients with American Society of Anesthesiologists (ASA) I and II scores
* patients over the age of 18

Exclusion Criteria:

* patients whose mouth and tongue mucosa integrity was degraded
* patients had a cognitive disorder
* patients had a neurological, renal, cardiac or pulmonary disorders that could affect the test results
* patients using psychoactive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
mouth dryness severity | Evaluation was made in the first 48 hours after surgery
  Numbered between 0-10 0: no dry mouth 10: very severe dry mouth Numerical rating scale (1-3 mild, 4-6 moderate, 7-10 severe) were used.
thirst severity | Evaluation was made in the first 48 hours after surgery
  Numbered between 0-10 0: no thirsty 10: very severe thirsty Numerical rating scale (1-3 mild, 4-6 moderate, 7-10 severe) were used.
saliva PH | Evaluation was made in the first 48 hours after surgery
  To measure the pH value, the patient's saliva sample were taken and simple PH test sticks were used and the PH value were determined according to the color changes on the PH test stick.
oral condition | Evaluation was made in the first 48 hours after surgery
  The Oral Health Assessment Tool were used. As the score on the scale increases, the oral condition worsens.

SECONDARY OUTCOMES:
patient satisfaction assessed by the VAS | It were evaluated at 48th hours postoperatively.
  VAS will be used, numbered between 0-10, 0: not satisfied at all, 10: very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Bediye Oztas, Phd, Principal Investigator — Ankara Medipol University
Locations (1):
- Gulhane Education and Training Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Oztas M, Oztas B. Effect of Spray Use on Mouth Dryness and Thirst of Patients Undergoing Major Abdominal Surgery: A Randomized Controlled Study. J Perianesth Nurs. 2022 Apr;37(2):214-220. doi: 10.1016/j.jopan.2021.04.018. Epub 2022 Feb 10. PMID 35153118